CLINICAL TRIAL: NCT01593501
Title: How Does Magnesium Status Influence Calcium Homeostasis?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC #2011-0547; R01AG028739-01A2 (NIH)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Magnesium Deficiency; Calcium Metabolism Disorders
Keywords: vitamin D; cholecalciferol; bone mineral density; Magnesium deficiency; Calcium metabolism disorders
MeSH Terms: conditions — Magnesium Deficiency; Calcium Metabolism Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose vitamin D (Active Comparator): 50,000 IU vitamin D3 every 15 days, with a loading dose of 50,000 IU per day for the first 15 days of an approximate 365-day treatment.
  Interventions: Dietary Supplement: vitamin D3
- Low dose vitamin D (Active Comparator): 800 IU vitamin D3 every day of an approximate 365-day treatment.
  Interventions: Dietary Supplement: vitamin D3
- Placebo (Placebo Comparator): A pill that looks like the low/high dose vitamin D pills, but contains no vitamin D. Given to preserve the double-blind nature of the study.
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3 — pharmaceutical grade D3
  Other Names: Cholecalciferol

SUMMARY:
The investigators aim to recruit 60 women who have agreed to participate in an existing randomized, double-blind, placebo-controlled trial (Treatment of Vitamin D Insufficiency, HSC 2009-0055). In this trial, the investigators propose to evaluate the associations between magnesium intake, magnesium stores, fractional magnesium absorption and calcium homeostasis. The investigators will stratify 60 subjects in the sub-study, ensuring that approximately 20 subjects are randomized into each treatment arm (placebo, low-dose and high-dose vitamin D). The investigators already assess calcium homeostasis throughout the study by measuring bone mineral density, fractional calcium absorption, serum and urine calcium levels, among other tests. In the sub-study of 60 women, the investigators will evaluate whether habitually higher magnesium intake increases or decreases fractional calcium absorption. The investigators will evaluate the interplay between magnesium stores, vitamin D levels and serum parathyroid hormone levels. The investigators will directly assess magnesium stores using serum magnesium and 24-hour urine magnesium levels, and will measure magnesium absorption using the dual stable isotope approach.

DETAILED DESCRIPTION:
Use of serum magnesium isotopes to measure fractional magnesium absorption Four day food diaries to assess magnesium intake Standard urine and serum chemistries for remaining labs as noted above

ELIGIBILITY:
Inclusion Criteria:

* participants eligible for the study "Treatment of vitamin D insufficiency" are eligible for participation in the current sub-study

Exclusion Criteria:

* identical to those covered in HSC #2009-0055

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the associations between magnesium intake, magnesium stores, fractional magnesium absorption and calcium homeostasis. | 0-12 months
  To evaluate relationships between magnesium intake and fractional magnesium absorption at baseline and 12 months, among 60 women participating in HSC Protocol 2009-0055, and to assess whether vitamin D therapy influences magnesium absorption among these women. We will also evaluate whether data collected from less than 72 hours of urine following tracer administration permits accurate assessment of fractional magnesium absorption.

SECONDARY OUTCOMES:
Does vitamin D therapy have a differential impact on calcium absorption that is dependent on magnesium stores? | 0-12 months
  To assess whether vitamin D therapy has a differential impact on calcium absorption, depending on magnesium stores. We will use data from all subjects participating in HSC Protocol 2009-0055 to evaluate whether magnesium status is a co-factor in the change in calcium absorption that occurs with vitamin D therapy.
Assessing relationships between magnesium status and bone mineral density. | 0-12 months
Evaluate how magnesium status impacts the relationship between vitamin D levels and parathyroid hormone levels. | 0-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hansen, M.D., M.S., Principal Investigator — University of Wisconsin-Madison, Department of Medicine, Division of Rheumatology
Locations (1):
- University of Wisconsin-Madison Hospital, Clinical Research Unit, Osteoporosis Research Center, Madison, Wisconsin, United States

REFERENCES:
- [Background] Hansen KE, Nabak AC, Johnson RE, Marvdashti S, Keuler NS, Shafer MM, Abrams SA. Isotope concentrations from 24-h urine and 3-h serum samples can be used to measure intestinal magnesium absorption in postmenopausal women. J Nutr. 2014 Apr;144(4):533-7. doi: 10.3945/jn.113.186767. Epub 2014 Feb 5. PMID 24500940